CLINICAL TRIAL: NCT07180589
Title: Advancing Assessment for Disorders of Consciousness (AADOC): Innovative Standards and Intelligent Diagnostic System Based on Multi-source Heterogeneous Information
Brief Title: Advancing Assessment for Disorders of Consciousness
Acronym: AADOC
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2024YFC3606901
Record Dates: First submitted 2025-08-25; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Disorders of Consciousness
Keywords: Disorders of consciousness; Prognostication
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past two decades, major progress has been made in detecting, predicting and promoting recovery of consciousness in patients with disorders of consciousness (DOC) caused by severe brain injuries. This study will aim to establish innovative standards and intelligent diagnostic system based on multi-source heterogeneous information including clinical signs, advanced neuroimaging and electrophysiological techniques, thus raising hope for more accurate diagnosis and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* age range: 18-80 years old; brain injury caused by various reasons, confirmed by clinical physical and chemical, neuroimaging (head MRI or CT) examination; Glasgow Coma Score (GCS)<12 points; modified Rankin Scale (mRS) score before the onset of the disease was less than 2 points; obtain informed consent from the patient's legal representative.

Exclusion Criteria:

* patients with significant skull defects; contraindications for electromagnetic related examinations and treatments, including the presence of metal materials in the body (such as pacemakers, dentures, steel nails, cochlear implants, etc.); patients with a history of epilepsy and clinical indications of epileptic seizures or epileptic discharges on electroencephalogram (EEG); women who are pregnant, breastfeeding, or have a positive pregnancy test upon admission; patients with an estimated survival period of less than 3 months due to various serious illnesses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with disorders of consciousness
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) at 1, 3, 6 and 12 months. | 12 months of disorders of consciousness onset
  Seven grades are set for scores of each item: 0-point (no disability), 1-point (no significant disability), 2-point (slight disability), 3-point (moderate disability), 4-point (moderate severe disability), 5-point (severe disability), and 6-point (death).

OTHER OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) at 1, 3, 6 and 12 months. | 12 months of disorders of consciousness onset
  The CRS-R scale consists of 23 hierarchically organized items divided into five functional subscales (auditory, visual, motor, oromotor/ verbal, communication) and an arousal scale. The sum of subscale values forms the total CRS-R score ranging between 0 and 23, with low values reflecting reflexive behavior and higher values indicating cognitively mediated behavior.
Glasgow Outcome Scale-Extended (GOSE) at 1, 3, 6 and 12 months. | 12 months of disorders of consciousness onset
  Eight grades are set for scores of each item: 1-point (dead), 2-point (vegetative state), 3-point (lower severe disability), 4-point (upper severe disability), 5-point (lower moderate disability), 6-point (upper moderate disability), 7-point (lower good recovery), and 8-point (upper good recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data and materials are available from the corresponding author upon reasonable request.